CLINICAL TRIAL: NCT06335485
Title: Digital Phenotyping to Monitor a CBT Pain Prevention Intervention for Women With Chronic Life Stress Undergoing Surgery
Brief Title: Cognitive Behavioral Therapy (CBT) Pain Prevention Intervention for Women Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Linda S Aglio, Anesthesiologist, Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020- P123456
Record Dates: First submitted 2023-06-23; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Back Pain; Cognitive Behavioral Therapy; Surgery
Keywords: Chronic stress; Elective spine surgery; Cognitive Behavioral Therapy; Digital Phenotyping; Fitbit tracker; Back Pain
MeSH Terms: conditions — Back Pain | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Patients are randomized to either the intervention group or general group, for the intervention group patients will be randomly assigned to attend 4 weekly online virtual CBT sessions that will provide information on stress and pain reduction techniques before surgery, and 2 sessions following patient surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT intervention group (Experimental): Participants will be asked to wear an activity tracker throughout the duration of the study. In addition, Participants will attend 4 weekly online virtual CBT sessions that will provide information on stress and pain reduction techniques before surgery, and 2 sessions following surgery.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- No CBT group (No Intervention): Participants will be asked to wear an activity tracker throughout the duration of the study.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Participants will attend 4 CBT sessions prior to surgery and 2 optional sessions after surgery.
  Arms: CBT intervention group

SUMMARY:
This study investigates a Cognitive Behavioral Therapy (CBT) intervention for women who are undergoing elective surgery. The objective is to provide a toolkit of stress management techniques to decrease pain and opioid use following surgery.

DETAILED DESCRIPTION:
The Investigators are doing this research to understand whether a pre-surgery virtual cognitive behavioral therapy (CBT) group intervention combined with an activity tracker can reduce pain and opioid use in women with chronic stress undergoing elective spine surgery.

Participants will be randomly divided in two groups and one of the groups will be invited to attend four weekly virtual CBT group sessions designed to improve reactions to stress, increase motivation for physical activity, develop tools for managing pain, and utilize mindfulness techniques. Two optional sessions will be available following surgery. Individuals randomized to usual care will not attend the online sessions but will continue to wear the activity tracker to provide information about their physical activity as well as the use of an App to track their pain and medication use.

The ultimate goal of this research is to enhance stress management and coping skills to help patients better manage pain after surgery and reduce their need for opioid medications.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Female Gender
3. Patients own a compatible smartphone (iPhone or Android) or tablet and can download the Fitbit app on their device
4. Planned elective spine surgery

Exclusion Criteria:

1. Cognitive impairment (judged to interfere with study participation)
2. Male gender
3. Non-English speaking
4. Pain conditions requiring urgent surgery
5. A diagnosis of cancer
6. A present psychiatric condition (e.g. DSM diagnosis of schizophrenia, delusional disorder, psychotic disorder or dissociative disorder) that would be judged to interfere with the study
7. Visual impairment or motor impairment that would interfere with study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Enrollment: 32 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating | At Baseline and weekly until 90 days.
  Research Subjects will be asked to rate their pain on a scale from 0-10.

SECONDARY OUTCOMES:
Pain Medication Usage | At Baseline and weekly until 90 days.
  Research Subjects will be asked to enter their pain medication usage prior to and after surgery. Medication type (opioid and non-opioid), dose, and quantity will entered into an online App that will be downloaded to the patients phone.
Activity Tracking (Digital Phenotyping) | At Baseline and weekly until 90 days.
  Investigators will quantify the amount of activity for each study subject (throughout the study up to 90 days) to establish the feasibility of collecting activity data on a wearable activity monitoring device before and after surgery. In addition, this activity data will be used to establish a digital phenotype by using statistical methods to identify clusters of women with similar recovery trajectories. Investigators will work to identify two distinct recovery patterns: optimal and slow.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States